CLINICAL TRIAL: NCT04767100
Title: Study of the Impact of a Social Telepresence Robot on Social Isolation and Loneliness of the Elderly at Home
Acronym: DOMIROB
Status: Completed | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00381-38
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Elderly People Living at Home; With an Internet Connection at Home
Keywords: Elderly people; Living at home; Internet connection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Social telepresence robot — Use of a social telepresence robot at home, during three months with the aim of reducing the feeling of loneliness and social isolation among the elderly.

SUMMARY:
The main purpose of this monocentric, prospective study is to measure the impact of the implementation of a robotic social telepresence tool, during three months at home, on the feeling of loneliness and social isolation of the elderly

DETAILED DESCRIPTION:
This non-interventional and prospective study offers elderly people living at home the opportunity to host a social telepresence robot, for a period of three months, with the aim of maintaining a link with those around them and discovering activities offered by professionals (cooking, yoga, visiting virtual museum, etc.) via a networking platform.

This study consists of questionnaires and score calculations, assessing their feeling of loneliness and how they accept the robot in their home.

Subjects will be interviewed one week before the robot arrives at their home, at the start of the study (when the robot arrives).

The follow-up is carried out by a neuropsychologist at 6, 12 and 24 weeks of presence at home.

Data measuring loneliness and social isolation, memory, patient interaction with the robot, their quality of life as well as their emotions will be collected using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged at least 65 and living at home in Ile-de-France
* Having expressed his non-opposition to his participation in the study
* Agreeing to host a social telepresence robot at home
* Having an internet connection at home

Exclusion Criteria:

* Subject aged under 65 or not living at home in Ile-de-France
* Having expressed his opposition to his participation in the study
* With moderate / major cognitive impairment (Mini-mental state examination (MMSE) <20)
* Placed under tutorship / curatorship
* Whose housing surface is insufficient for reception and robot movements

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly subjects living at home, volunteers, divided into 6 groups of 10 people. This represents a simultaneous implementation of 10 robots at home.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Measuring subjective feelings of loneliness as well as feelings of social isolation according the UCLA Loneliness Scale | 24 weeks
Measuring the perception of social support according Multidimensional Scale of Perceived Social Support | 24 weeks

SECONDARY OUTCOMES:
Measuring the perceived usability of the robot's software according the System Usability Scale | 24 weeks
Measuring technology acceptance according ALMERE questionnaire | 12 weeks
Assessment of the impact of health according 12-Item Short Form Survey (SF-12) scale | 24 weeks
Assessment of depressive state according Geriatric Depression Scale | 24 weeks
Assessment positive and negative affect according the Positive Affect Negative Affect Scale (PANAS) | 24 weeks
Assessment of the psycho-social impact of the device technology on the lives of users according The Psychosocial Impact of Assistive Devices Scales (PIADS) | 12 weeks
Measuring the dimensions of the telepresence according Telepresence Temple Presence Inventory (TPI) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie RIGAUD, MD PhD, Study Chair — Living Lab Department, Broca Hospital
Locations (1):
- Living Lab Department, Broca Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Isabet B, Rigaud AS, Li W, Pino M. Telepresence Robot Intervention to Reduce Loneliness and Social Isolation in Older Adults Living at Home (Project DOMIROB): Protocol for a Clinical Nonrandomized Study. JMIR Res Protoc. 2022 Oct 31;11(10):e40528. doi: 10.2196/40528. PMID 36315231